CLINICAL TRIAL: NCT00663377
Title: Losartan Improved Insulin Resistance and Decreased Inflammatory Cytokines in Patients With Chronic Heart Failure Treated With Angiotensin Converting Enzyme Inhibitors
Brief Title: Effects of Losartan on Insulin Resistance in Patients With Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tottori University Hospital (Other)
Responsible Party: Kazuhide Ogino, Center for Clinical Residency Program, Tottori University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: #656
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Heart Failure
Keywords: Heart Failure; Insulin Resistance; Losartan; ACE inhibitor; Inflammatory cytokine
MeSH Terms: conditions — Heart Failure; Insulin Resistance | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: losartan — losartan 50-100mg for 16 weeks

SUMMARY:
The purpose of this study is to evaluate the effects of losartan, an ARB, on glucose metabolism and inflammatory cytokines in CHF patients treated with ACE inhibitors.

DETAILED DESCRIPTION:
Chronic heart failure (CHF) is associated with marked insulin resistance, characterized by both fasting and stimulated hyperinsulinemia. Furthermore, insulin resistance is a predictor of CHF and associated with more severe disease and a worse prognosis in patients with CHF. In CHF patients, therefore, insulin resistance is not merely a function of adiposity and may have implications in the pathophysiology of CHF disease progression. Angiotensin II negatively modulates insulin-mediated actions by regulating multiple levels of the insulin signaling cascade such as the insulin receptor, IRS, and PI3-kinase. Furthermore, both ACE inhibitors and angiotensin II receptor blockers (ARB) improve glycemic status not only in patients with type II diabetes but also in patients with hypertension and the metabolic syndrome. On the other hand, it is well known that some cytokines, such as TNF-α, are involved with pathophysiology of insulin resistance and CHF. However, it is still unclear whether the ARB improves insulin resistance in CHF patients already treated with ACE inhibitors and whether there is the relationship between insulin resistance and inflammatory cytokines in CHF patients already treated with ACE inhibitors. Therefore, the purpose of this study is to evaluate the effects of losartan, an ARB, on glucose metabolism and inflammatory cytokines in CHF patients treated with ACE inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* chronic stable heart failure

Exclusion Criteria:

* renal dysfunction or under treatment with antidiabetic agents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2006-04; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
insulin resistance | 16 weeks

SECONDARY OUTCOMES:
inflammatory cytokines | 16 weeks

REFERENCES:
- [Derived] Ogino K, Kato M, Furuse Y, Kinugasa Y, Kaetsu Y, Mizuta E, Sugihara S, Ishida K, Yanagihara K, Hisatome I, Shigemasa C. Addition of losartan to angiotensin-converting enzyme inhibitors improves insulin resistance in patients with chronic heart failure treated without beta-blockers. Circ J. 2010 Nov;74(11):2346-52. doi: 10.1253/circj.cj-10-0395. Epub 2010 Sep 4. PMID 20827028